CLINICAL TRIAL: NCT03448484
Title: Programme Effectiveness of an Integrated Programme to Reduce Maternal and Child Malnutrition in Kenya: Cluster Randomized, Parallel-group, Prospective, Follow-up Effectiveness Study in Children 6-35 Months of Age at Recruitment
Brief Title: Cluster Randomized, Parallel-group, Prospective, Follow-up Effectiveness Study in Kenyan Children 6-35 Months
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fabian Rohner (Other)
Collaborators: One Acre Fund (Unknown); Children's Investment Fund Foundation (Other)
Responsible Party: Sponsor-Investigator, Fabian Rohner, President, GroundWork
Organization: GroundWork (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: GW_1AF_KenEff_U5
Record Dates: First submitted 2018-02-22; First posted 2018-02-28 (Actual); Last update posted 2021-07-28 (Actual); Status verified 2021-07

CONDITIONS: Stunting
MeSH Terms: conditions — Growth Disorders | interventions — Methods

STUDY DESIGN:
Intervention Model Description: Cluster Randomized, Parallel-group, Prospective, Follow-up Effectiveness Study
Who Masked: Outcomes Assessor
Masking Description: The nature of the intervention package compared to the control package prevents a double-blind study design and thus, only the outcome assessors (data collectors) and the study statistician can be blinded to the group assignment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Intervention (agriculture-focused package + nutrition-sensitive and nutrition-specific interventions=integrated package)
  Interventions: Dietary Supplement: Intervention (integrated package)
- Control (Other): Control (agriculture-focused package)
  Interventions: Other: Control

INTERVENTIONS:
Dietary Supplement: Intervention (integrated package) — Provided to all intervention households:
  * Soap (for daily hand washing)
  * Chlorine solution (for daily drinking water treatment)
  * 8 birds of chicken (child consumes 1 egg/day)
  * Vegetable seeds (red onion, indigenous managu and sukuma)
  * Monthly trainings to all farmers on nutrition and WASH
  * Micronutrient powder (MixMe, 1g sachet every third day)
  * Oral rehydration solution (ORS) + zinc (to be used to treat acute diarrhoea: 20 mg zinc tablets; ORS sachets (10.3 g/sachet))
  All families in the intervention group will receive the same agriculture-focused package (see section 'control intervention' below) as those in the control group.
  Arms: Intervention
Other: Control — Active control: The families living in the control clusters will receive the agriculture-focused package that is already in place in all participating clusters through the 1AF programme. The control intervention is the same for study 1 and study 2. This agriculture-focused package consists of:
  * Agricultural training (every 2 weeks on average) for all
  * Free to enrol for the following products on credit:
    * Compost boosters
    * Cook stoves
    * Seeds (onions, maize, indigenous greens, beans)
    * Maize storage bags
    * Drying tarps
    * Trees
    * Solar lights
    * Fertilizer
    * Actellic dust (insecticide)
    * Re-usable sanitary pads
  Arms: Control

SUMMARY:
Malnutrition is a public health problem in Kenya, with 26% of children under-five years of age stunted, and 26% of pre-school children, 26% of women of reproductive age and 42% of pregnant women being anaemic, respectively. Agriculture is the main source of income, food and nutrients for the majority of rural families in Sub-Saharan Africa including Kenya. Most farmers are smallholders and are vulnerable to poor nutrition. Thus far, programmes have mostly focused on increasing yields and household income, but not on improving nutritional status. One Acre Fund (1AF) has over the past 10 years successfully introduced an agriculture programme to smallholder farmers in Western Kenya focusing on improving harvest. 1AF is therefore well placed to transform an existing and successful agriculture programme into the world's largest 'nutrition network' for farmers, and it is the hope that a partnership between Children's Investment Fund Foundation (CIFF) and 1AF will create a strong voice for nutrition within the agriculture sector. The project aims to use an integrated programme by introducing nutrition-sensitive (improved water, sanitation and hygiene (WASH): e.g. soap for hand washing) and nutrition-specific (e.g. micronutrient supplements) components to 1AF's agricultural programme.

The impact of such an integrated programme will be assessed in a cluster-randomized intervention study in children 6-35 months at recruitment comparing one group receiving the integrated intervention to another group receiving the agricultural intervention (already in place).

DETAILED DESCRIPTION:
Background/introduction:

Malnutrition, and particularly malnutrition in children under 5 years of age, remains a public health problem in many areas of the world [1]. A diet low in diversity and micronutrient density is one contributing factor while a second factor is poor water, sanitation and hygiene (WASH) practices often leading to diseases such as persistent diarrhoea and resulting in morbidity and mortality in children under 5 years of age. According to the WHO World Health Statistics 2017 that are monitoring health in order to reach the Sustainable Development Goals (SDGs) [2] including data from between 2006 and 2015, the global under 5 mortality rate per 1000 live birth is 42.5 and is clearly highest in the African Region with 81.3 while in Kenya it is lower than the African average with 49.4. The picture is similar for maternal mortality with 216 per 100,000 live births globally but with the highest in the African region with 542 and 510 in Kenya.

The statistics also look at several WASH indicators. The mortality rate attributed to exposure to unsafe WASH services per 100,000 populations is clearly highest in the African region with a burden of 43.1, while the global burden is at 12.4, and with Kenya slightly below the African burden with 32.5. In line with this, two additional WASH indicators demonstrate the poor status in the African region. The use of improved drinking water source is lowest in the African region with 68%, while globally 91% use an improved source and in all the other WHO regions it is over 90%. Kenya is slightly below the African average with 63% using an improved drinking water source. Looking at sanitation the use of improved sanitation is lowest in the African region with only 32% and is similar at the Kenyan level with 30% while globally 68% use improved sanitation. The most recent Kenya Demographic and Health Survey in 2014 estimates that only about a third of households in Kenya have washing places at their homes [3]. Also, nationally, three out of four households share toilets with other households or have unimproved toilets (open defecation, open latrines, etc.). Malnutrition is specifically covered in SDG Target 2.2 (By end 2030, end all forms of malnutrition, including achieving, by 2025, the internationally agreed targets on stunting and wasting in children under 5 years of age, and address the nutritional needs of adolescent girls, pregnant and lactating women and older persons). The WHO statistics indicate a worldwide problem with 22.9% of children under 5 years of age stunted and 7.7% wasted. While the Africa Region (33.5% and 7.4%)) together with the South-East-Asia Region (33.8% and 15.3)) have the highest stunting and wasting prevalence, respectively, the prevalence in Kenya is below the Africa average with 26.0% stunted and only 4% wasted.

Agriculture is the main source of income, food and nutrients for the majority of rural families in Sub-Saharan Africa including Kenya. Most rural families in Sub-Saharan Africa are smallholder farmers, and rely on agricultural produce for income and direct consumption. Despite the fact that these households are food producers, research has shown that rural farming households are typically net food consumers and are more vulnerable to malnutrition [4]. Decades of investments in the agriculture sector have focused on improving yields and income but have notably failed to improve the nutrition status of farming families and their children [5]. Since 2006, One Acre Fund (1AF) has been providing a bundle of services and agricultural inputs to smallholder farmers using a model where farmers take loans to pay for inputs and services received. The core service bundle includes environmentally appropriate seed and fertilizer, physical delivery of inputs, training, and small loans. 1AF currently reaches 445,000 farming households in Kenya, Burundi, Rwanda, Tanzania, Malawi, and Uganda. Kenya was 1AF's first country of operation and their activities will soon cover all of Western and Nyanza Provinces, which are the primary food-producing regions and hold one third of Kenya's population. The most recent 1AF report impressively shows the increasing number of farm families served, the Dollar gain in farmer impact and the close to 100% farmer repayment rate of credits for seeds and fertilizers [6].

In partnership with the Children's Investment Fund Foundation (CIFF), 1AF aims to introduce nutrition-sensitive and nutrition-specific components into the services offered to smallholder farmer households. The nutrition-specific interventions consist of providing MNPs (Micronutrient Powders) to children 6-59 months of age. These nutritional supplements are recommended by WHO in areas where micronutrient deficiencies and malnutrition are prevalent [7,8]. In order to increase protein consumption, chicken birds will be provided to households. Households will also be provided with seeds for red onion and indigenous greens. Further, children will be provided with oral rehydration salts (ORS) and zinc supplements as recommended by WHO and UNICEF for the treatment of acute diarrhoea [9]. Lastly, some WASH related interventions will also be provided, such as training sessions, soap for hand washing and chlorine for drinking water treatment.

To test the incorporation of nutrition services in 1AF's agricultural programme, pilot projects in western Kenya will be conducted between 2017 and 2020. The dietary diversity, food frequency and subsequently, a minimum acceptably dietary quality for young children are lower in the Western Province than for the national average. Further, the number of households with washing places is lower and diarrhoea prevalence is slightly higher compared to the national average [3].

In order to monitor and evaluate 1AF's programmes, a cluster-randomized, parallel-group, prospective, follow-up effectiveness study in children 6-35 months of age at recruitment that spans over 2 years will be conducted in the Western Province of Kenya.

Clusters will be randomly assigned to either have the regular 1AF agricultural intervention package (already in place in all clusters participating in the study and therefore called control) or the integrated intervention package that on top of the agricultural package consists of nutrition-specific (such as providing additional micronutrients) and nutrition-sensitive (such as providing soap for hand washing) interventions. The impact on malnutrition and programmatic 'success' will be evaluated.

Objective/hypothesis:

While the primary purpose is to longitudinally compare the changes of growth between the intervention and control group, the programmatic aspects such as adherence to and coverage of the intervention package and possible links to changes in dietary patterns and ultimately linear growth will also be evaluated.

As such, the research hypothesis is as follows: Linear growth in children between 6-59 months of age will improve after the provision of agricultural services, nutritionally enhanced and WASH products and diversified crops as well as nutrition and WASH training over the period of 2 years when compared to the control group provided only with agricultural services.

Study design:

The general study design is a cluster-randomized, parallel-group, prospective, follow-up effectiveness study over a period of 2 years comparing 2 groups of children 6-35 months of age at recruitment:

1. Intervention group: All selected households with children 6-35 months of age at recruitment will receive MNP (1 sachet every three days per child) and ORS along with zinc (20 mg/day) for treatment of acute diarrhoea. The households will also be provided with soap, chlorine solution, poultry (8 chickens at start of intervention), and seeds for red onion and indigenous greens (March 2018 and March 2019). The products will be accompanied by monthly nutrition and WASH trainings. The products and trainings will be provided free of charge. Additionally, all households will receive the agricultural package as in the control group.
2. Control group: All households will be provided with agricultural training (every 2 weeks on average) for free. In addition, households can also enrol for the following products on credit: compost booster, cook stoves, seeds (onions, maize, indigenous greens, beans), maize storage bags, drying tarps, trees, solar lights, fertilizer, actellic dust (insecticide), re-usable sanitary pads.

We anticipate recruiting 2,000 (1,000 in each group) children 6-35 months of age into the study. Children will be recruited from 100 clusters (randomly assigned to intervention or control) that will be drawn from Lugari district in Kakamega County located in the Western Province of Kenya.

Questionnaire based and anthropometric data will be collected in 3 rounds at a central place in walking distance from participant's homes one year apart from each other (Table 4). The following information will be collected in round 1 (baseline assessment prior to the actual start of intervention distribution):

* Age
* Height and weight
* Household demographics/characteristics and caregiver's education
* Dietary diversity, breastfeeding and infant and young children feeding (IYCF) practices
* WASH practices
* Child morbidity In rounds 2 and 3, information on dietary diversity, breastfeeding and IYCF practices, WASH practices and child morbidity will be collected again. Additionally, changes in adherence and coverage of the intervention package as well as unintended outcomes (e.g. reduction of exclusive breastfeeding due to premature introduction of complementary foods) will be assessed.

References:

1. Development Initiatives (2017) Global Nutrition Report 2017: Nourishing the SDGs. Bristol, UK: Development Initiatives.
2. WHO (2017) World Health Statistics 2017: Monitoring health for the SDGs, Sustainable Development Goals. http://apps.who.int/iris/bitstream/10665/255336/1/9789241565486-eng.pdf?ua=1: Geneva: World Health Organization.
3. DHS (2015) Kenya Demographic and Health Survey 2014. http://dhsprogram.com/pubs/pdf/FR308/FR308.pdf: Kenya National Bureau of Statistics, Ministry of Health, Nationla AIDS Control Council, Kenya Medical Research Institute, National Council for Population and Development, The DHS Program, ICF International.
4. Senbanjo IO, Olayiwola IO, Afolabi WA, Senbanjo OC (2013) Maternal and child under-nutrition in rural and urban communities of Lagos state, Nigeria: the relationship and risk factors. BMC Res Notes 6: 286.
5. Fanzo J (2014) Strengthening the engagement of food and health systems to improve nutrition security: Synthesis and overview of approaches to address malnutrition. Global Food Security 3: 183-192.
6. 1AF (2016) One Acre Fund- Annual Report 2016. https://www.oneacrefund.org/uploads/all-files/2016_AnnualReport_r1.pdf: One Acre Fund.
7. WHO (2007) Preventing and controlling micronutrient deficiencies in populations affected by an emergency. http://www.who.int/nutrition/publications/micronutrients/WHO_WFP_UNICEFstatement.pdf: World Health Organisation, World Food Programme, UNICEF
8. WHO (2016) WHO guideline: Use of multiple micronutrient powders for point- of- use fortification of foods consumed by infants and young children aged 6- 23 months and children aged 2-12 years. http://apps.who.int/iris/bitstream/10665/252540/1/9789241549943-eng.pdf?ua=1: Geneva: World Health Organization.
9. WHO/UNICEF (2004) Clinical management of acute diarrhoea. http://apps.who.int/iris/bitstream/10665/68627/1/WHO_FCH_CAH_04.7.pdf: World Health Organization, UNICEF.

ELIGIBILITY:
Inclusion Criteria:

* Children 6-35 months of age at recruitment
* Caregiver providing written informed consent to participate

Exclusion Criteria:

* Family does not intend to stay within the study area for at least the following 24 months
* Visible severe disease

Ages: 6 Months to 35 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1927 (Actual)
Dates: Start 2018-03-12 (Actual); Primary Completion 2020-07-01 (Actual); Study Completion 2020-10-01 (Actual)

PRIMARY OUTCOMES:
Stunting and length/height-for-age z-score | 2 years
  Change in length-for-age z-score (LAZ) over the course of the two years programme activity

SECONDARY OUTCOMES:
Nutrient density | 2 years
  Change in nutrient density due to increased consumption of MNPs and improved crops
Dietary diversity | 2 years
  Change in dietary diversity due to increased adherence to adequate child feeding practices
Breastfeeding | 2 years
  Proportion of children still breastfed
WASH behaviour | 2 years
  Proportion of households with soap and water available

CONTACTS AND LOCATIONS:
Overall Officials: Rita Wegmüller, Principal Investigator — GroundWork
Locations (1):
- One Acre Fund, Kakamega, Kenya

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Adu-Afarwuah S, Lartey A, Okronipa H, Ashorn P, Peerson JM, Arimond M, Ashorn U, Zeilani M, Vosti S, Dewey KG. Small-quantity, lipid-based nutrient supplements provided to women during pregnancy and 6 mo postpartum and to their infants from 6 mo of age increase the mean attained length of 18-mo-old children in semi-urban Ghana: a randomized controlled trial. Am J Clin Nutr. 2016 Sep;104(3):797-808. doi: 10.3945/ajcn.116.134692. Epub 2016 Aug 17. PMID 27534634
- [Background] Ashorn P, Alho L, Ashorn U, Cheung YB, Dewey KG, Gondwe A, Harjunmaa U, Lartey A, Phiri N, Phiri TE, Vosti SA, Zeilani M, Maleta K. Supplementation of Maternal Diets during Pregnancy and for 6 Months Postpartum and Infant Diets Thereafter with Small-Quantity Lipid-Based Nutrient Supplements Does Not Promote Child Growth by 18 Months of Age in Rural Malawi: A Randomized Controlled Trial. J Nutr. 2015 Jun;145(6):1345-53. doi: 10.3945/jn.114.207225. Epub 2015 Apr 29. PMID 25926413
- [Background] Matias SL, Mridha MK, Tofail F, Arnold CD, Khan MS, Siddiqui Z, Ullah MB, Dewey KG. Home fortification during the first 1000 d improves child development in Bangladesh: a cluster-randomized effectiveness trial. Am J Clin Nutr. 2017 Apr;105(4):958-969. doi: 10.3945/ajcn.116.150318. Epub 2017 Mar 8. PMID 28275128
- [Derived] Wegmuller R, Musau K, Vergari L, Custer E, Anyango H, Donkor WES, Kiprotich M, Siegal K, Petry N, Wirth JP, Lewycka S, Woodruff BA, Rohner F. Effectiveness of an integrated agriculture, nutrition-specific, and nutrition-sensitive program on child growth in Western Kenya: a cluster-randomized controlled trial. Am J Clin Nutr. 2022 Aug 4;116(2):446-459. doi: 10.1093/ajcn/nqac098. PMID 35421217

DOCUMENTS (1):
  • Study Protocol (2018-01-15): https://cdn.clinicaltrials.gov/large-docs/84/NCT03448484/Prot_000.pdf